CLINICAL TRIAL: NCT01656928
Title: Effects of a Pre-school-based Nutritional Intervention on Children's Eating Behavior and Anthropometric Parameters: a Cluster-randomized Trial
Brief Title: Effects of a Pre-school-based Nutritional Intervention on Children's Eating Behavior and Anthropometric Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Joachim E. Fischer, Professor Dr. med. MSc, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRTLasti_nutr_kiga
Record Dates: First submitted 2012-07-27; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting-list control (Other): Allocation to waiting-list Control. Receives intervention 6 months later.
  Interventions: Behavioral: preschool-based nutritional intervention
- Intervention (Active Comparator): Allocation to intervention. Directly starts with nutritional intervention.
  Interventions: Behavioral: preschool-based nutritional intervention

INTERVENTIONS:
Behavioral: preschool-based nutritional intervention — 6-month intervention administered once weekly by a nutrition expert consisting of joint meal preparation and activities for children and parents such as tasting and preparing nutritious, fresh foods.
  Other Names: Nutritional Module of program "Komm mit in das gesunde Boot"

SUMMARY:
This study assesses the impact of a nutritional intervention aimed at reducing childhood overweight in German preschoolers.

DETAILED DESCRIPTION:
Objective: To assess the impact of a nutritional intervention aimed at reducing childhood overweight in German preschoolers.

Design: Using a cluster-randomized study design with waiting-list controls, we test a six-month intervention administered once weekly by a nutritional expert consisting of joint meal preparation and activities for children and parents like tasting and preparing nutritious, fresh foods. At baseline, six and twelve months, a parent-completed questionnaire assesses fruit and vegetable intake (primary outcomes) and water and sugared drink consumption (other outcomes). Direct measurement assessed BMI, percentage body fat (skin fold thicknesses) and waist-to-height-ratio. An intention-to-treat analysis used random effects panel regression models to assess the intervention effect, adjusted for each child's age, gender, immigrant background and maternal education.

Setting: 18 Preschools from three south German regions. Subjects: Healthy children from three to seven years of age.

ELIGIBILITY:
Inclusion Criteria:

* Pre-schools were eligible to participate in the study if they were located in one of three predefined regions and had applied to participate in the nutritional intervention module of a state-sponsored health promotion programme 'Komm mit in das gesunde Boot' ('Come aboard the health boat'), with at least fifteen children participating.
* Healthy children in eligible preschools

Exclusion Criteria:

* Age under 3 years or above 7 years
* Serious health problems
* Genetic conditions
* Metabolic diseases
* Acute infectious diseases

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in Fruit- and vegetable consumption | 0, 6, 12 months
  Before intervention (0 months), at the end of intervention (6 months), six months after intervention (12 months)

SECONDARY OUTCOMES:
Change in Body Mass Index | 0, 6, and 12 months
  Before intervention (0 months), at the end of intervention (6 months), six months after intervention (12 months)
Change in Percent body fat | 0, 6 and 12 months
  Before intervention (0 months), at the end of intervention (6 months), six months after intervention (12 months)
Change in waist-to-height ratio | 0, 6 and 12 months
  Before intervention (0 months), at the end of intervention (6 months), six months after intervention (12 months)

OTHER OUTCOMES:
Change in water consumption; Change in juice consumption | 0, 6 and 12 months
  Before intervention (0 months), at the end of intervention (6 months), six months after intervention (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E Fischer, Professor Dr.med. MSc, Principal Investigator — University of Heidelberg, Mannheim Institute of Pubic Health
Locations (1):
- Mannheim Institute of Public Health, University of Heidelberg, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] De Bock F, Breitenstein L, Fischer JE. Positive impact of a pre-school-based nutritional intervention on children's fruit and vegetable intake: results of a cluster-randomized trial. Public Health Nutr. 2012 Mar;15(3):466-75. doi: 10.1017/S136898001100200X. Epub 2011 Aug 23. PMID 21859516